CLINICAL TRIAL: NCT06222216
Title: The Effect of Chilled Needle on the Development of Pain and Ecchymosis in Subcutaneous Injection in Adults: A Prospective, Randomized Controlled Study
Brief Title: The Effect of Chilled Needle on the Development of Pain and Ecchymosis in Subcutaneous Injection in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali Kaplan, Assist. Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Ali KAPLAN - Kayseri U
Record Dates: First submitted 2024-01-11; First posted 2024-01-24 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Pain; Ecchymosis; A Randomized Controlled Trial; Subcutaneous Injections
MeSH Terms: conditions — Pain; Ecchymosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Chilled Needle): (Experimental): Before subcutaneous injection, 26G sterile disposable needles will be kept in the cooling compartment of the refrigerator for at least 24 hours. Immediately before SC injection, the needle will be removed from the refrigerator, placed in the ice box and placed next to the patient's bed. The needle temperature will be kept at 0-2 degrees Celsius in the ice box and controlled using an LCD digital thermometer. If Enoxaparin Sodium is in the ready injector, the drug in the injector will be drawn into the injector suitable for 1 cc SC injection application without loss of dose. The needle of the prepared syringe will be replaced with a cooled needle. Afterwards, the injection will be made in the designated area (outer side of the upper arm) in accordance with the SC injection procedure steps. After the injection, the patient's pain assessment will be made and marked on the ILC, and ecchymosis assessment will be made after 24, 48 and 72 hours.
  Interventions: Other: Chilled Needle
- Control Group: (Active Comparator): SC injection will be administered to the control group in accordance with the clinical routine. No different procedure will be applied. Injection will be performed with a needle at room temperature without any instrument or procedure in accordance with the SC injection protocol. After the injection, the patient's pain assessment will be made and marked on the SCI, and ecchymosis assessment will be made after 24, 48 and 72 hours.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Chilled Needle — Before subcutaneous injection, 26G sterile disposable needles will be kept in the refrigerated compartment of the refrigerator for at least 24 hours. Immediately before SC injection, the needle will be removed from the refrigerator, placed in the ice box and placed next to the patient's bed. The needle temperature will be kept at 0-2 degrees Celsius in the ice box and controlled using an LCD digital thermometer. If Enoxaparin Sodium is in the ready injector, the drug in the injector will be drawn into the injector suitable for 1 cc SC injection application without loss of dose. The needle of the prepared syringe will be replaced with a cooled needle. Afterwards, the injection will be made in the designated area (outer side of the upper arm) in accordance with the SC injection procedure steps. After the injection, the patient's pain assessment will be made and marked on the ILC, and ecchymosis assessment will be made after 24, 48 and 72 hours.
  Arms: Intervention Group (Chilled Needle):
Other: Control Group — SC injection will be administered to the control group in accordance with the clinical routine. No different action will be applied. The injection will be made in accordance with the SC injection protocol with a needle at room temperature, without applying any tools or procedures. After the injection, the patient's pain will be evaluated and marked on the VAS, and ecchymosis will be evaluated after 24, 48 and 72 hours.
  Arms: Control Group:

SUMMARY:
Subcutaneous (SC) injection applications are the process of administering the drug to the loose connective tissue under the skin and is one of the most frequently applied parenteral drug administration methods among nursing practices. SC injections, which are frequently performed by nurses, often result in complications such as hematoma, ecchymosis and pain at the injection site. Although the field of healthcare is developing day by day, injection applications can still be painful and uncomfortable. These procedures increase the individual's stress levels before the procedure, causing them to experience fear and anxiety and reducing patient satisfaction. This may cause the application to fail or be repeated. Many nonpharmacological methods are applied to prevent or reduce these local side effects in subcutaneous injection applications. Cold application is accepted as an effective and easy-to-use method for SC injection. Cold application may also constrict peripheral blood vessels, reducing blood flow to the tissue and thus preventing ecchymosis.

When the national and international literature is examined, there are studies using cold application to reduce pain and ecchymosis due to SC injection in adults. This study aimed to evaluate the effectiveness of cold injection, which is considered an alternative to cold therapy, in reducing pain and ecchymosis due to SC injection application. No study has been found in the literature evaluating the effectiveness of cold injection in preventing pain and ecchymosis due to SC injection application. Therefore, it is thought that this study will make a significant contribution to the literature and create a simple, comfortable and cost-free innovation. Preparation and use of cold injection is simple, easy and comfortable. It is anticipated that patients will be able to easily follow the procedure steps during the procedure. Therefore, this study aimed to examine the effect of the cooled needle on the development of pain and ecchymosis in SC injection application in adults.

DETAILED DESCRIPTION:
Subcutaneous (SC) injection applications are the process of administering the drug to the loose connective tissue under the skin and is one of the most frequently applied parenteral drug administration methods among nursing practices. SC injections, which are frequently performed by nurses, often result in complications such as hematoma, ecchymosis and pain at the injection site. Although the field of healthcare is developing day by day, injection applications can still be painful and uncomfortable. These procedures increase the individual's stress levels before the procedure, causing them to experience fear and anxiety and reducing patient satisfaction. This may cause the application to fail or be repeated. Factors affecting pain and ecchymosis caused by subcutaneous injection include injection time, injection site, drug injected, dose injected, and needle size. Many nonpharmacological methods are applied to prevent or reduce these local side effects in subcutaneous injection applications. Cold application is accepted as an effective and easy-to-use method for SC injection. Cold application may also constrict peripheral blood vessels, reducing blood flow to the tissue and thus preventing ecchymosis.

When the national and international literature is examined, there are studies using cold application to reduce pain and ecchymosis due to SC injection in adults. This study aimed to evaluate the effectiveness of cold injection, which is considered an alternative to cold therapy, in reducing pain and ecchymosis due to SC injection application. No study has been found in the literature evaluating the effectiveness of cold injection in preventing pain and ecchymosis due to SC injection application. Therefore, it is thought that this study will make a significant contribution to the literature and create a simple, comfortable and cost-free innovation. Preparation and use of cold injection is simple, easy and comfortable. It is anticipated that patients will be able to easily follow the procedure steps during the procedure. Therefore, this study aimed to examine the effect of the cooled needle on the development of pain and ecchymosis in SC injection application in adults.

The research will be conducted as a randomized controlled, experimental clinical trial. The population of the research will consist of patients who applied to Erciyes University Health Application and Research Center General Surgery Service between the dates of the study. As a result of the analysis, it was decided to include a total of 60 people in the sample of the research. In collecting research data, the Case Report Form consisting of the Individual Introduction Form, Visual Comparison Scale and Ecchymosis Tracking Chart, created by the researchers by scanning the relevant literature, will be used. The data obtained in the research will be analyzed using the SPSS 24.0 program. Care will be taken to comply with ethical principles at every stage of the research. Before starting the application, an Academic Board Decision, ethics committee approval from the ERÜ Faculty of Medicine Ethics Committee and institutional permission from the ERÜ Health Application and Research Center will be obtained. Participants will first be explained the purpose of the research, given information about the research, and their written consent (Informed Volunteer Consent Form) will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Able to speak and understand Turkish,
2. Those between the ages of 18-65,
3. Oriented to place and time,
4. Having no vision or hearing problems,
5. Not using psychiatric medication due to any psychiatric disease,
6. Not using central nervous system medication,
7. Not using narcotic analgesics,
8. Having a Visual Comparison Scale pain score of zero at the time of application,
9. Those who have not had SC injection in the last month,
10. Low molecular weight heparin therapy is ordered (Enoxaparin Sodium 1*4000 IU),
11. Having an average pressure pain threshold of 8-16 pounds (Lb) with the Baseline Algometer device,
12. Has normal platelet, INR, and aPTT values,
13. Individuals who volunteer to participate in the study and sign the written voluntary consent form will be included in the research.

Exclusion Criteria:

1. Vital signs not within the reference range,
2. Those with signs of phlebitis, scar tissue, dermatitis, incision and infection in the area where the intervention will be performed,
3. Having had a mastectomy,
4. Patients who declare that they are addicted to alcohol and drugs will not be included in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Individual Introduction Form | 6 months
  The form prepared by the researcher by examining the relevant literature; individuals' age, gender, marital status, etc. It consists of 7 questions that include socio-demographic characteristics such as. The individual identification form will be filled out by the researcher by meeting individuals face to face.
Visual Comparison Scale | 6 months
  The Visual Comparison Scale is a scale used to measure pain intensity. It is used to convert the pain value that cannot be measured numerically into numerical form. Two extreme definitions of the pain parameter are written at both ends of a 100 mm line, and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line, placing a dot, or pointing. It is a 100 mm (10 cm) ruler that can be used horizontally and vertically, with "painlessness" written on one end and "most severe pain possible" on the other end. "0 mm" means no pain, and "100 mm" means the most severe pain. The individual indicates the intensity of pain he feels on this ruler. Pain intensity score measurements will be evaluated in mm.
Octoberosis Tracking Chart | 6 months
  It is a form developed by researchers to track the development of ecchymosis in patients after subcutaneous injection, in which the date and time of SC injection and the ecchymosis at 24, 48, and 72 hours after injection are recorded.
  In the project, an acetate pen will be used to measure ecchymosis in the injection area. In the literature, color changes smaller than 2 mm2 are not considered ecchymosis. Based on this information, in this study, color change smaller than 2 mm will be categorized as "no ecchymosis" and color change 2 mm and above will be categorized as "ecchymosis present".

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical faculty hospital, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No